CLINICAL TRIAL: NCT00366093
Title: The Efficacy of Eszopiclone 3 mg Compared to Placebo in the Treatment of Insomnia Secondary to Perimenopause or Menopause
Brief Title: Study of Eszopiclone Compared to Placebo in the Treatment of Insomnia Secondary to Perimenopause/Menopause
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sumitomo Pharma America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 190-054
Record Dates: First submitted 2006-08-17; First posted 2006-08-18 (Estimated); Last update posted 2012-02-22 (Estimated); Status verified 2012-02

CONDITIONS: Insomnia
Keywords: Menopause; Perimenopause
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Eszopiclone

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): eszopiclone 3 mg
  Interventions: Drug: Eszopiclone
- 2 (Placebo Comparator): Placebo tablet
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Eszopiclone — eszopiclone 3 mg
  Other Names: Lunesta; S-zopiclone
  Arms: 1
Drug: Placebo — placebo tablet
  Arms: 2

SUMMARY:
To demonstrate improved subjective sleep in women with insomnia secondary to perimenopause or menopause following treatment with 3 mg of eszopiclone.

DETAILED DESCRIPTION:
A multicenter, randomized, double-blind, placebo-controlled, parallel-group study of eszopiclone 3 mg in women with insomnia secondary to perimenopause or menopause. Eligible subjects will be randomized to either eszopiclone 3 mg or placebo nightly for four weeks. This study was previously posted by Sepracor Inc. In October 2009, Sepracor Inc. was acquired by Dainippon Sumitomo Pharma., and in October 2010, Sepracor Inc's name was changed to Sunovion Pharmaceuticals Inc.

ELIGIBILITY:
Inclusion Criteria

* Subject must understand the purpose of the study and be willing to adhere to the study schedule and procedures described in this protocol.
* Subject must be between the ages of 40 and 60 years, inclusive, on the day of signing consent.
* Subject must have perimenopausal or menopausal signs and symptoms.
* Subject must report SL of >45 minutes and <6 hours of TST at least three times a week over the previous month and symptoms of insomnia must post date onset of perimenopausal or menopausal symptoms.
* Subject's physical exam must show no clinically significant abnormal findings (other than insomnia and menopause symptoms) at screening.

Exclusion Criteria

* Subject has history of circadian rhythm disorder, or travels across >3 time zones on a regular basis.
* Female subject is pregnant, lactating or within 6-months post partum.
* Subject has a history of drug or alcohol abuse or dependence in the past 2 years or positive urine drug test at screening .
* Subject has unstable medical abnormality, or unstable chronic disease; or history of significant cardiac, renal, or hepatic disease, seizure disorder, or current or past acute suicidal tendencies.
* Subject has participated in any investigational drug study within 30 days prior to screening or plans to participate in another investigational drug study during participation in this study.
* Subject is taking hormone replacement therapy or an hormonal contraceptive, and has not been on a stable dose for a minimum of 60 days prior to study start.
* Subject is known to be seropositive for HIV.
* Subject has a disorder or history of a condition (e.g., malabsorption, gastrointestinal surgery) that may interfere with drug absorption distribution, metabolism, or excretion.
* Subject has a history of malignancy within 5 years, or current malignancy, except for non-melanoma skin cancer.
* Subject has a diagnosis of any psychiatric disorder as identified by a psychiatric screening questionnaire.
* Subject has any primary diagnosis (personality disorder or mental retardation) that would impact the investigator's ability to evaluate the safety or efficacy of the study medication.
* Subject has difficulties in sleep initiation or maintenance associated with other known primary sleep disorders [e.g. sleep apnea, restless leg syndrome (RLS), or periodic leg movement syndrome (PLMS)], or has any condition that may affect sleep (e.g., chronic pain, urinary incontinence, etc.).
* Subject has used any drugs known or suspected to affect hepatic or renal clearance capacity within a period of 30 days prior to screening.
* Subject reports consumption of more than two alcoholic beverages daily, 14 or more alcoholic beverages weekly, or five or more alcoholic beverages on any given day.
* Subject is a rotating or third/night shift worker.
* Subject is a staff member or relative of a staff member.
* Subject is experiencing symptoms of premature menopause or surgical menopause.
* Subject has discontinued hormone replacement therapy or a hormonal contraceptive, and has not been off treatment for a minimum of 60 days prior to study start.
* Subject has been on hormone replacement therapy or hormonal contraceptives for greater then one year.

Ages: 40 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 410 (Actual)
Dates: Start 2004-02; Primary Completion 2005-01 (Actual); Study Completion 2005-01 (Actual)

PRIMARY OUTCOMES:
mean subjective SL | Week 1

SECONDARY OUTCOMES:
mean subjective WASO | Week 1
Mean subjective SL | Weeks 2, 3, 4
Mean subjective WASO | Weeks 2, 3, 4
Mean subjective TST | Weeks 1, 2, 3, 4
Mean number of awakenings | Weeks 1, 2, 3, 4
Sleep quality and depth | Weeks 1, 2, 3, and 4
Daytime alertness | Weeks 1, 2, 3, and 4
Ability to concentrate | Weeks 1, 2, 3, and 4
Physical well-being | Weeks 1, 2, 3, and 4
Ability to function | Weeks 1, 2, 3, and 4
Mean subjective number of nocturnal awakenings due to hot flashes | Weeks 1, 2, 3, and 4
Mean number of hot flashes per day | Weeks 1, 2, 3, and 4
Mean number of nocturnal hot flashes per night | Weeks 1, 2, 3, and 4
Mean severity of hot flashes | Weeks 1, 2, 3, and 4
ESS score | Weeks 2 and 4
ISI score | Weeks 2 and 4
GCS score | Weeks 2 and 4
SDS score | Week 4
MenQOL score | Week 4
MADRS score | Week 4
Physician Global Assessment | Week 4
withdrawal effects will be assessed for the ISI, ESS, MADRS, MenQOL, Greene Climacteric Scale, Sheehan Disability Scale, and Physician Global Assessment. | Week 5

CONTACTS AND LOCATIONS:
Locations (51):
- United States (51):
  - Mobile, Alabama
  - San Diego, California
  - Denver, Colorado
  - Newington, Connecticut
  - Aventura, Florida
  - Clearwater, Florida
  - Fort Meyers, Florida
  - Gainesville, Florida
  - Melbourne, Florida
  - Miami, Florida
  - Naples, Florida
  - New Port Richey, Florida
  - Pembroke Pines, Florida
  - Tampa, Florida
  - West Palm Beach, Florida
  - Atlanta, Georgia
  - Savannah, Georgia
  - Arlington Heights, Illinois
  - Champaign, Illinois
  - Chicago, Illinois
  - Lexington, Kentucky
  - Louisville, Kentucky
  - Boston, Massachusetts
  - Brockton, Massachusetts
  - Ann Arbor, Michigan
  - St Louis, Missouri
  - Lincoln, Nebraska
  - Reno, Nevada
  - Rochester, New York
  - Cary, North Carolina
  - Raleigh, North Carolina
  - Winston-Salem, North Carolina
  - Cleveland, Ohio
  - Dayton, Ohio
  - Mentor, Ohio
  - Oklahoma City, Oklahoma
  - Medford, Oregon
  - Erie, Pennsylvania
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Warwick, Rhode Island
  - Columbia, South Carolina
  - Cordova, Tennessee
  - Houston, Texas
  - Irving, Texas
  - Sandy City, Utah
  - Richmond, Virginia
  - Renton, Washington
  - Seatle, Washington
  - Spokane, Washington
  - Tacoma, Washington

REFERENCES:
- [Derived] Soares CN, Joffe H, Rubens R, Caron J, Roth T, Cohen L. Eszopiclone in patients with insomnia during perimenopause and early postmenopause: a randomized controlled trial. Obstet Gynecol. 2006 Dec;108(6):1402-10. doi: 10.1097/01.AOG.0000245449.97365.97. PMID 17138773